CLINICAL TRIAL: NCT06981780
Title: Accuracy of the Change in Femoral Artery Doppler Indices as Novel Predictors to Successful Caudal Block in Pediatric Patients a Prospective Observational Study
Brief Title: Change in Femoral Artery Doppler to Predict Successful Caudal Block
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Adolf Helmy, Lecturer of anesthesia and critical care, Cairo University
Other Study IDs: Doppler and caudal block
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Caudal Block
Keywords: Femoral artery Doppler; Pulsatility index; Caudal block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Femoral artery Doppler: Each patient will be examined using femoral artery Doppler at 3 timepoints
  Interventions: Device: Femoral artery Doppler

INTERVENTIONS:
Device: Femoral artery Doppler — An experienced operator will conduct femoral artery examination for the change in Doppler indices namely pulsatility index, resisitive index, and waveform morphology

SUMMARY:
The ideal method to predict successful caudal block is still lacking. We hypothesized that the change in femoral artery Doppler indices could accurately predict successful caudal block

DETAILED DESCRIPTION:
after institutional research ethics committee approval and obtaining informed consent from each participant. an experienced operator will examine the femoral artery using pulsed wave Doppler at baseline and 15 and 30 minutes after caudal block adminestration

ELIGIBILITY:
Inclusion Criteria:

* ASA1 or 2 lower abdominal or lower limb surgery

Exclusion Criteria:

* allergy to bupivacaine parental refusal coagulopathy inability to obtain adequate femoral artery views

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients undergoing abdominal or lower limb surgery under general anesthesia combined with caudal block
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2025-05-20 (Actual); Primary Completion 2025-08-20 (Actual); Study Completion 2025-08-21 (Actual)

PRIMARY OUTCOMES:
Accuracy of Change in pulsatility index (PI) to predict successful caudal block | baseline and 15 minutes after the block
  The change in PI measured at baseline and 15 minutes after the block

SECONDARY OUTCOMES:
Accuracy of the change in resistive index to successful caudal block | baseline and 15 minutes
  The change in RI at baseline and 15 minutes after the block
accuracy of change in waveform morphology to predict successful caudal block | baseline and 15 minutes after the block
  The change in femoral artery waveform from triphasic to a monophasic wave

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data regarding this study will be available from the corresponding author upon reasonable request

REFERENCES:
- [Background] Xu Z, Zhang J, Shen H, Zheng J. Assessment of pulse oximeter perfusion index in pediatric caudal block under basal ketamine anesthesia. ScientificWorldJournal. 2013 Sep 19;2013:183493. doi: 10.1155/2013/183493. eCollection 2013. PMID 24174910
- [Background] Adolf Helmy M, Mansour M, Magdy Milad L, Mohammed Aboelregal E, Magdy Youssef M. Change in femoral artery pulsatility index as a novel predictor of post-spinal anesthesia hypotension in adult patients undergoing infra-umbilical surgeries: A prospective observational study. Anaesth Crit Care Pain Med. 2025 Apr;44(2):101482. doi: 10.1016/j.accpm.2025.101482. Epub 2025 Jan 21. No abstract available. PMID 39848332
- [Background] Kim ES, Sharma AM, Scissons R, Dawson D, Eberhardt RT, Gerhard-Herman M, Hughes JP, Knight S, Marie Kupinski A, Mahe G, Neumyer M, Poe P, Shugart R, Wennberg P, Williams DM, Zierler RE. Interpretation of peripheral arterial and venous Doppler waveforms: A consensus statement from the Society for Vascular Medicine and Society for Vascular Ultrasound. Vasc Med. 2020 Oct;25(5):484-506. doi: 10.1177/1358863X20937665. Epub 2020 Jul 15. PMID 32667274
- [Background] Boretsky KR, Camelo C, Waisel DB, Falciola V, Sullivan C, Brusseau E, Eastburn E, Gomez-Moraz A, Luckanavanich W. Confirmation of success rate of landmark-based caudal blockade in children using ultrasound: A prospective analysis. Paediatr Anaesth. 2020 Jun;30(6):671-675. doi: 10.1111/pan.13865. PMID 32267040
- [Background] Kao SC, Lin CS. Caudal Epidural Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:9217145. doi: 10.1155/2017/9217145. Epub 2017 Feb 26. PMID 28337460